CLINICAL TRIAL: NCT06936657
Title: Intervention Effects of Optimized Carbohydrate Diet in Patients With Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Huating, Professor, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-018
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimized carbohydrate diet-washout-conventional diabetes diet (Experimental): Group that starts with the optimized carbohydrate diet
  Interventions: Other: optimized carbohydrate diet; Other: conventional diabetes diet
- conventional diabetes diet-washout-optimized carbohydrate diet (Experimental): Group that starts with the conventional diabetes diet
  Interventions: Other: optimized carbohydrate diet; Other: conventional diabetes diet

INTERVENTIONS:
Other: optimized carbohydrate diet — In this dietary pattern, 50-60% of total energy is derived from carbohydrates, 15-20% from protein, and 25-30% from fat. Among the carbohydrates, resistant starch (RS) constitutes 15-20% of daily starch intake (around 40 g/day), slowly digestible starch (SDS) 5%, rapidly digestible starch (RDS) 75-80%, with dietary fiber at 20-40g per 1000 kcal and free sugars contributing less than 5% of total energy.
Other: conventional diabetes diet — In this dietary pattern, 50-60% of total energy is derived from carbohydrates, 15-20% from protein, and 25-30% from fat. Among the carbohydrates, resistant starch (RS) constitutes 5% of daily starch intake, slowly digestible starch (SDS) 5%, rapidly digestible starch (RDS) 90%, with dietary fiber at 14g per 1000 kcal and free sugars contributing less than 5% of total energy.

SUMMARY:
This study is a multi-center, randomized, crossover investigator-initiated trial conducted at Shanghai Sixth People's Hospital and other centers. Each participant will undergo two 12-week dietary intervention phases, separated by a 6-week washout, for a total study duration of 30 weeks. Participants will be randomly assigned in a 1:1 ratio to one of two intervention order: (1) optimized carbohydrate diet-washout-conventional diabetes diet, or (2) conventional diabetes diet-washout-optimized carbohydrate diet. The optimized carbohydrate diet is a modified diet with adjusted carbohydrate composition and proportions, while the conventional diabetes diet adheres to an energy-matched protocol in accordance with diabetes dietary guidelines. The study aims to explore the effects of the optimized carbohydrate diet on blood glucose control and glucose metabolism in patients with type 2 diabetes, and to systematically assess its impact on cognitive function and a range of physiological and psychological indicators (such as depression, anxiety, appetite, sleep, bowel habits and others).

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with type 2 diabetes according to the ADA diagnostic criteria
2. HbA1c ≥ 7% and < 9%
3. Antidiabetic medication has been stable for at least 3 months before recruitment
4. Aged 35-70 years
5. Signed the informed consent form

Exclusion Criteria:

1. Treatment with insulin
2. Treatment with GLP-1 receptor agonists or DPP-4 inhibitors
3. Occurrence of diabetic ketoacidosis, lactic acidosis, hyperosmolar coma, or recurrent severe hypoglycemia within the past year
4. Having one or more severe chronic diabetic complications, including advanced diabetic retinopathy, macroalbuminuria (urine albumin-to-creatinine ratio ≥300 mg/g), or impaired renal function (eGFR ≤60 ml/min/1.73 m²)
5. Presence of cardiovascular events (e.g., myocardial infarction, stent placement, unstable angina, heart failure, cardiac dysfunction) or cerebrovascular diseases (e.g., intracerebral hemorrhage, ischemic stroke) within the past 6 months
6. Diagnosis of acute or chronic gastrointestinal diseases (e.g., ulcers), hyperthyroidism or hypothyroidism, uncontrolled hypertension, active malignancy not in remission, or other life-threatening diseases
7. Recent use of antibiotics, probiotics, or prebiotics within the past 3 weeks or need for long-term use
8. Unstable medication regimen or use of prescription medications affecting metabolism (e.g., thyroid hormones, glucocorticoids)
9. Pregnancy, breastfeeding, or planning pregnancy
10. Presence of a pacemaker or metal implants, claustrophobia, or other contraindications to fMRI
11. Psychiatric disorders impairing cooperation
12. Expected poor compliance
13. Current or recent (within 4 weeks prior to study initiation) participation in other clinical trials

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in the average incremental area under the curve (iAUC) of postprandial blood glucose over 3 hours | -2, 0, 10, 16, 18 and 28 weeks
  Average incremental area under the curve (iAUC) of postprandial blood glucose over 3 hours will be measured at -2, 0, 10, 16, 18, and 28 weeks using the continuous glucose monitoring system.

SECONDARY OUTCOMES:
Change in other parameters of Continuous Glucose Monitoring | -2, 0, 10, 16, 18 and 28 weeks
  Other parameters of Continuous Glucose Monitoring, including Time in Range (TIR), Time Above Range (TAR), Time Below Range (TBR), Mean Glucose, Glucose Variability, Glycemic Excursions, Area Under the Curve (AUC), and other relevant metrics, will be assessed at -2, 0, 10, 16, 18, and 28 weeks.
Change in HbA1c | Baseline, 12, 18 and 30 weeks
  HbA1c will be measured at baseline, 12, 18 and 30 weeks. HbA1c will be expressed in mmol/mol.
Change in insulin sensitivity | Baseline, 12, 18 and 30 weeks
  Insulin sensitivity will be assessed at baseline, 12, 18 and 30 weeks.
Change in other clinical biochemical indicators | Baseline, 4, 8, 12, 18, 22, 26 and 30 weeks
  Other clinical biochemical indicators will be measured at baseline, 4, 8, 12, 18, 22, 26 and 30 weeks.
Change in blood glucose | Baseline, 4, 8, 12, 18, 22, 26 and 30 weeks
  Fasting blood glucose will be measured at baseline, 4, 8, 12, 18, 22, 26 and 30 weeks. During meal tolerance test (MTT) at baseline, 12, 18 and 30 weeks, blood glucose at 0, 30, 60, 90, 120 minutes will be measured. Glucose concentration will be expressed in mmol/L
Change in insulin and C peptide secretion | Baseline, 4, 8, 12, 18, 22, 26 and 30 weeks
  Fasting insulin and C peptide concentration will be assessed at baseline, 4, 8, 12, 18, 22, 26 and 30 weeks. During meal tolerance test (MTT) at baseline, 12, 18 and 30 weeks, insulin and C peptide concentration at 0, 30, 60, 90, 120 minutes will be measured. Insulin concentration will be expressed in uU/ml. C peptide concentration will be expressed in ng/ml.
Change in anthropometry and body composition parameters | Baseline, 4, 8, 12, 18, 22, 26 and 30 weeks
  Anthropometry and body composition parameters will be measured at baseline, 4, 8, 12, 18, 22, 26 and 30 weeks.
Change in cognitive function and behavioral performance | Baseline, 12, 18 and 30 weeks
  Cognitive function changes will be assessed using questionnaires (including the Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA, Beijing version), Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), Trail Making Test, Stroop Color and Word Test, and others) at baseline, 12 18, and 30 weeks. Behavioral performance will be assessed using N-back and other paradigms at baseline, 12, 18, and 30 weeks.
  In addition, subgroups within the two arms will undergo fMRI to assess cognitive function at baseline, 12 18, and 30 weeks.
Change in appetite | Baseline, 12, 18 and 30 weeks
  Appetite will be measured by visual analog scales (VAS) and other relevant scales, and will be assessed at baseline, 12, 18, and 30 weeks.
Change in emotion | Baseline, 12, 18 and 30 weeks
  Emotion will be measured using the PHQ-9 depression screening scale, the Problem Areas in Diabetes (PAID) questionnaire, and other relevant scales at baseline, 12, 18, and 30 weeks.
Change in sleep quality | Baseline, 12, 18 and 30 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) questionnaire and other methods at baseline, 12, 18, and 30 weeks.
Change in bowel habits | Baseline, 12, 18 and 30 weeks
  Bowel habits will be assessed using the Bristol Stool Form Scale (BSFS; range: 1-7, with higher scores indicating looser stools) and other relevant scales at baseline, 12, 18, and 30 weeks.
Change in cardiopulmonary exercise testing performance | Baseline, 12, 18 and 30 weeks
  Cardiopulmonary exercise testing performance will be conducted at baseline, 12, 18 and 30 weeks.
Change in blood lipid profiles | Baseline, 4, 8, 12, 18, 22, 26 and 30 weeks
  Blood lipid profiles will be measured at baseline, 4, 8, 12, 18, 22, 26 and 30 weeks.

OTHER OUTCOMES:
Change in the iAUC of postprandial blood glucose over 3 hours after each meal | -2, 0, 10, 16, 18 and 28 weeks
  The iAUC of postprandial blood glucose over 3 hours after each meal in patients with type 2 diabetes will be measured at -2, 0, 10, 16, 18, and 28 weeks using the continuous glucose monitoring system.
Change in hepatic fat content | Baseline, 12, 18 and 30 weeks
  Hepatic fat content will be assessed by Fibroscan at baseline, 12, 18 and 30 weeks.
Change in the levels of cytokines | Baseline, 12, 18 and 30 weeks
  The levels of cytokines, including FGF21, adiponectin, A-FABP, LCN2, and others, will be assessed using Enzyme-Linked Immunosorbent Assay (ELISA) and other methods at baseline, 12, 18, and 30 weeks.
Change in immunologic function | Baseline, 12, 18 and 30 weeks
  The immunologic function will be assessed through isolation and analysis of peripheral blood mononuclear cells at baseline, 12, 18, and 30 weeks.
Change in appetite-related hormones | Baseline, 12, 18 and 30 weeks
  Concentration of appetite-related hormones (e.g., ghrelin, PYY, GLP-1 and others) will be measured at baseline, 12, 18, and 30 weeks.
Change in multi-omics | Baseline, 4, 8, 12, 18, 22, 26 and 30 weeks
  Multi-omics research, including metagenomic sequencing, metabolomics analysis, proteomics, lipidomics, genomics, etc., will be assessed at baseline, 4, 8, 12, 18, 22, 26 and 30 weeks.

REFERENCES:
- [Derived] Lu Y, Zhang R, Yang J, Liu D, Wu Q, Long X, Cheng D, Guo J, Li Q, Zhang Y, Kang P, Wang Q, Gao X, Zeng R, Zhang M, Fang Q, Jia W, Ni Y, Li H. Intervention effects of optimised carbohydrate diet in patients with type 2 diabetes: study protocol for a randomised controlled crossover trial. BMJ Open. 2025 Oct 7;15(10):e106756. doi: 10.1136/bmjopen-2025-106756. PMID 41062131